CLINICAL TRIAL: NCT02620956
Title: Aerosol Deposition in Asthmatic Obese Women Using Heliox: A Randomized, Crossover, Controlled Clinical Trial Study
Brief Title: Aerosol Deposition in Asthmatic Obese Women Using Heliox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jacqueline de Melo Barcelar (Other)
Responsible Party: Sponsor-Investigator, Jacqueline de Melo Barcelar, principal investigator, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 669.576.484-00
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Obese; Asthma
MeSH Terms: conditions — Obesity; Asthma | interventions — heliox; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- obese nebulizer (Active Comparator): would be used to inhale an aerosol with technetium labeled diethylenetriaminepente-acetic acid (99mTc - DTPA) with an activity of 1 mCi in a total dose volume with normal saline of 2,5 ml and heliox using a vibrating mesh inhaler.
  Interventions: Other: nebulizing with heliox and oxygen
- asthmatic obese nebulizer (Experimental): would be used to inhale an aerosol with technetium labeled diethylenetriaminepente-acetic acid (99mTc - DTPA) with an activity of 1 mCi in a total dose volume with normal saline of 2,5 ml and heliox using a vibrating mesh inhaler.
  Interventions: Other: nebulizing with heliox and oxygen

INTERVENTIONS:
Other: nebulizing with heliox and oxygen — Mesh Nebulizer with heliox and oxygen. In order to determine the sequence of the gas associated with the inhaled a randomization was performed, sequence 1- first oxygen and second heliox (80:20) or sequence 2- first heliox (80:20) and secondy oxygen.

SUMMARY:
BACKGROUND: The aim of this study was to assess pulmonary deposition and distribution of radio-aerosol in obese and normal women, using 2-D planar scintigraphy. METHODS: after inhaling an aerosol of technetium labeled diethylenetriamine penteacetic acid (99mTc - DTPA) with an activity of 1 mCi in a total dose volume with normal saline of 2,5 ml using a vibrating mesh inhaler.

DETAILED DESCRIPTION:
BACKGROUND: Obese asthmatics are difficult to treat effectively, worse asthma control, and do not respond as well to standard therapy as lean asthmatic. Medical aerosols an important route of drug delivery in asthma, but narrowing in the airway cause by the obesity, can provoke turbulence and the effectiveness of the treatment could be compromise.

AIM: To assess pulmonary deposition, distribution of radio-aerosol and analyze upper way dimension in obese and normal weight women, using 2-D planar scintigraphyand and computed tomography. METHODS: 20 obese women, 10 asthmatics and 10 non-asthmatics took part of the first part of the study. Anthropometric and clinical assessments were carried out, than lung function was performed. After randomization of the sequence of gas (sequence 1- oxygen and heliox; sequence 2-heliox and heliox) that would be used to inhale an aerosol with technetium labeled diethylenetriamine penteacetic acid (99mTc - DTPA) with an activity of 1 mCi in a total dose volume with normal saline of 2,5 ml using a vibrating mesh inhaler. All patients inhaled two times with one week of washout between then to eliminate risk of residual trace radiation and to avoid the possibility of bias.

ELIGIBILITY:
Inclusion Criteria:

* Were women with Body mass Index (BMI) ≥30kg/m2 for obese and BMI =18.5 - 24.9 kg/m2 for the control group
* Age between 18 to 60 years old
* With and without moderate to severe asthma
* Positive response to bronchodilator (improvement in FEV1 and/or FVC of at least 12% and 200ml).

Exclusion Criteria:

* Were women with active pulmonary disease other than asthma
* Neuromuscular diseases
* Smokers and those incapable of performing procedures were excluded.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Aerosol deposition in pulmonary compartments | two days

SECONDARY OUTCOMES:
Aerosol deposition in vertical and horizontal gradient | two days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital the Federal University of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Darquenne C, Prisk GK. Aerosol deposition in the human respiratory tract breathing air and 80:20 heliox. J Aerosol Med. 2004 Fall;17(3):278-85. doi: 10.1089/jam.2004.17.278. PMID 15625820
- [Background] Hess DR, Fink JB, Venkataraman ST, Kim IK, Myers TR, Tano BD. The history and physics of heliox. Respir Care. 2006 Jun;51(6):608-12. PMID 16723037
- [Background] Fink JB. Opportunities and risks of using heliox in your clinical practice. Respir Care. 2006 Jun;51(6):651-60. PMID 16723042
- [Background] Niimi A, Matsumoto H, Amitani R, Nakano Y, Mishima M, Minakuchi M, Nishimura K, Itoh H, Izumi T. Airway wall thickness in asthma assessed by computed tomography. Relation to clinical indices. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1518-23. doi: 10.1164/ajrccm.162.4.9909044. PMID 11029371